CLINICAL TRIAL: NCT00688493
Title: A Double-blind, Randomized, Four-period Crossover Study to Assess the Effects of Single Oral Dose Dapagliflozin Administration on QTc Interval Compared to Placebo, Using AVELOX™ (Moxifloxacin) as a Positive Control, in Healthy Male Volunteers Age 18 to 45 Years
Brief Title: Effects of Single Oral Dose Dapagliflozin QT Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: D1690C00001
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
Keywords: QT; Healthy volunteers
MeSH Terms: interventions — dapagliflozin; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 20 mg single dose of dapagliflozin (Experimental): 20 mg dapagliflozin
  Interventions: Drug: Dapagliflozin; Drug: Moxifloxacin; Drug: Placebo to match moxifloxacin and dapagliflozin
- 150 mg single dose of dapagliflozin2 (Experimental): 150 mg dapagliflozin
  Interventions: Drug: Dapagliflozin; Drug: Moxifloxacin; Drug: Placebo to match moxifloxacin and dapagliflozin
- 400 mg single dose of moxifloxacin (Active Comparator): Moxifloxacin
  Interventions: Drug: Dapagliflozin; Drug: Moxifloxacin; Drug: Placebo to match moxifloxacin and dapagliflozin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Dapagliflozin; Drug: Moxifloxacin; Drug: Placebo to match moxifloxacin and dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — 3 x 50 mg tablets, single oral dose
Drug: Dapagliflozin — 2 x 10 mg capsules, single oral dose
Drug: Moxifloxacin — Overencapsulated 400 mg capsule, single oral dose
  Other Names: Avelox™
Drug: Placebo to match moxifloxacin and dapagliflozin — Overencapsulated 400 mg capsule, single oral dose

SUMMARY:
The main purpose of this study is to examine the effect of dapagliflozin on electronic measures of heart beats in healthy males

ELIGIBILITY:
Inclusion Criteria:

* Healthy males age 18 to 45 years of age, who are not currently taking any medications
* Normal screening results including a physical examination, laboratory tests, heart rate, blood pressure, and ECG (electronic measure of the heart)

Exclusion Criteria:

* No personal or family history of significant heart problems
* No use of over the counter medications within 7 days of the study
* No use of prescription medicaiton within 1 month of the study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-07; Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Electronic measures of heart beats | ECGs (electronic measures of the heart) are taken at scheduled times during the 3 days after receiving each dose of study medication

SECONDARY OUTCOMES:
Blood levels of dapagliflozin following single 20 mg and 150 mg doses in healthy volunteers | At scheduled times during the 3 day periods following dosing during each of the 4 study periods
Safety and tolerability of dapagliflozin | Screening through completion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Carlson, MD, Study Director — AstraZeneca; Ronald Goldwater, MD, Principal Investigator — Parexel
Locations (1):
- Research Site, Baltimore, Maryland, United States